CLINICAL TRIAL: NCT00014339
Title: A Randomized, Phase III, Placebo-Controlled Multicenter Study to Demonstrate the Effectiveness and Safety of the Combination Enzyme Tablet (Wobe-Mugos E) as Adjuvant Therapy to Standard of Care Treatment in Patients With Stages II or III Multiple Myeloma
Brief Title: Chemotherapy With or Without Wobe-Mugos E in Treating Patients With Stage II or Stage III Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medsearch (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068535; MEDSEARCH-MU-699-501; MUCOS-MU-699-501
Record Dates: First submitted 2001-04-10; First posted 2004-02-26 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — chymotrypsin, papain, trypsin drug combination; Melphalan; Prednisone

INTERVENTIONS:
Drug: Wobe-Mugos E
Drug: melphalan
Drug: prednisone
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Enzyme products such as Wobe-Mugos E may help to reduce the side effects of multiple myeloma therapy. It is not yet known if chemotherapy is more effective with or without Wobe-Mugos E in treating multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy with or without Wobe-Mugos E in treating patients who have stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the long-term survival of patients with chemotherapy-naive stage II or III multiple myeloma treated with standard melphalan and prednisone with or without adjuvant Wobe-Mugos E. II. Compare the effect of these two regimens on the reduction of the side effects from chemotherapy in these patients, using 2 quality of life questionnaires. III. Compare the effect of these two regimens on tumor response rate and new metastasis development in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive oral melphalan and oral prednisone on days 1-4. Patients also receive adjuvant enzyme therapy with oral Wobe-Mugos E 3 times daily beginning prior to or on day 1 of the first course of chemotherapy. Arm II: Patients receive melphalan and prednisone as in arm I. Patients also receive an oral placebo 3 times daily as in arm I. Treatment continues for a minimum of 12 months to up to 4 years in the absence of unacceptable toxicity. Patients continue on melphalan and prednisone on a 4-week course until achieving maximum response or plateau phase and then receive 2 additional courses of therapy. Quality of life is assessed at baseline; at 1, 3, and 6 months and every 6 months for up to 4 years during study; and then at end of study. Patients are followed for survival for 1 month after completing the study and all patients receive the enzyme product.

PROJECTED ACCRUAL: A total of 250 patients (125 per treatment arm) will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage II or III multiple myeloma by bone marrow biopsy or aspiration Previously untreated with chemotherapy Melphalan and prednisone as only choice of standard treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 1 year Hematopoietic: WBC at least 2,000/mm3 Absolute neutrophil count at least 1,000/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT or SGPT no greater than 3 times upper limit of normal (ULN) PT or PTT no greater than 1.2 times ULN Renal: Creatinine no greater than 2.0 mg/dL (if stage IIA or IIIA) Creatinine greater than 2.0 mg/dL (if stage IIB or IIIB) Cardiovascular: No myocardial infarction within the past 6 months No congestive heart failure Other: No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell cancer or carcinoma in situ of the cervix No other disease, psychiatric condition, or substance abuse that would preclude study No serious non-malignant disease, including uncontrolled infection or peptic ulcer disease HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior transplantation or stem cell therapy No concurrent interferon therapy during initial melphalan and prednisone regimen Chemotherapy: See Disease Characteristics Concurrent other chemotherapy allowed if disease progression on study therapy Endocrine therapy: Not specified Radiotherapy: No more than 6 months since prior localized radiotherapy Concurrent localized radiotherapy allowed Surgery: Not specified Other: At least 30 days since prior investigational drug therapy Concurrent bisphosphonates for bone disease required No other concurrent enzyme preparation (including over the counter or nutraceutical preparations) No concurrent participation in other clinical study No concurrent anticoagulant therapy unless medically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Hildegard Frichtel, MD, Study Chair — Medsearch
Locations (19):
- United States (19):
  - Southwest Clinical Research, Incorporated, Phoenix, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Southwest Cancer Care, Poway, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oncology Radiation Associates, Miami, Florida
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Indiana Community Cancer Care, Inc., Indianapolis, Indiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - Oncology Hematology Associates of Kansas City, Kansas City, Missouri
  - HemOnCare, P.C., Brooklyn, New York
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - West Clinic, P.C., Memphis, Tennessee
  - Hematology Oncology Northwest, P.C., Tacoma, Washington